CLINICAL TRIAL: NCT03839485
Title: Endodontic Treatment of Primary Teeth With Guedes-Pinto Paste Without Antibiotic: Randomized Non-inferiority Clinical Trial
Brief Title: Endodontic Treatment of Primary Teeth With Guedes-Pinto Paste Without Antibiotic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fausto Medeiros Mendes, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FouspPGP
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Pulp Disorder
Keywords: pulpectomy; primary teeth; root canal filling materials
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Pulpectomy; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both materials will be packed in identical and opaque syringes, identified only with letters (A and B). The codes will be revealed only at the end of the study. Neither the professional who will be performing the treatment, nor the patient or the evaluator, who will perform the exams at follow-up times, will know which of the two materials of choice were selected for each tooth, characterizing the study as triple-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pasta Guedes-Pinto (Active Comparator): Endodontic treatment using Guedes-Pinto Paste
  Interventions: Drug: Endodontic treatment using Guedes-Pinto Paste
- Pasta Guedes-Pinto without antibiotic (Experimental): Endodontic using Guedes-Pinto paste without antibiotic
  Interventions: Drug: Endodontic using Guedes-Pinto Paste without antibiotic

INTERVENTIONS:
Drug: Endodontic treatment using Guedes-Pinto Paste — Dental procedure in which the entire pulp chamber is removed from the crown and roots of a tooth and the root filling material Guedes-Pinto paste is applied
  Other Names: Pulpectomy with Guedes-Pinto paste
  Arms: Pasta Guedes-Pinto
Drug: Endodontic using Guedes-Pinto Paste without antibiotic — Dental procedure in which the entire pulp chamber is removed from the crown and roots of a tooth and the root filling material Guedes-Pinto paste without antibiotic is applied
  Other Names: Pulpectomy with Guedes-Pinto paste without antibiotic
  Arms: Pasta Guedes-Pinto without antibiotic

SUMMARY:
The pulp therapy in primary teeth is still necessary even with all odontopediatrics evolution in prevention and minimal intervention, aiming to keep the tooth free of inflammation or infection and in a functional state until its exfoliation. Several materials are used as filling paste of primary teeth. In Brazil, the Guedes-Pinto Paste (PGP), an association of iodofórmio, camphorated paramonochlorophenol, prednisolone and rifamycin, has been widely used for some decades. However, current Brazilian legislation has made it difficult to commercialize antibiotics, which has made it difficult to obtain the ointment that is the association between prednisolone and rifamycin. Therefore, the objective of this clinical trial will be to test PGP without rifamycin in the pulpectomy of primary teeth, and to compare it with the treatment performed with conventional PGP.

DETAILED DESCRIPTION:
A randomized triple-blind non-inferiority clinical study with two parallel arms, with a 12-month follow-up, will be performed. The experimental group will be PGP formulated without the antibiotic, while the control group is the conventional PGP, containing rifamycin. The conventional pulpectomy will be performed using manual files, performing the instrumentation aided by Endo-PTC and 1% sodium hypochlorite. At the end of the instrumentation, just before the obturation, the groups will be drawn, with the strategy of randomization in permuted blocks and stratified by the initial condition of the tooth (with or without periapical lesion). The main outcome will be the clinical and radiographic success of endodontic treatment after 12 months. Patients who seek the dental service of the municipality and require endodontic treatment will be invited to participate in the study. The data will be statistically analyzed using the statistical package Stata 12.0 (Stata Corporation, College Station, TX, USA). The longevity of the treatments will be evaluated by estimating survival rates using the Kaplan-Meier method. The differences between survival rates according to the type of endodontic treatment proposed will be analyzed through the Log-rank test.

ELIGIBILITY:
Inclusion Criteria:

* Primary molar teeth with necessity of endodontic treatment.
* Patients whose parents or guardians consent to their participation in the study

Exclusion Criteria:

* Systemic health problems, congenital facial deformities, facial tumors or syndromes
* Teeth presenting one of the following:

  * Resorption of more than 2/3 of the root
  * Destruction of the crypt of the permanent successor
  * Pulp chamber floor drilling.
  * Presence of internal resorption

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Success or failure of treatment | 1 year
  The success or failure of endodontic treatments evaluated by the time spent in the tooth arch in clinical conditions of normality. Clinical criteria for determining success are: absence of fistula, absence of painful symptoms and pathological absence of adequate mobility and gingival contour. Radiographically, the success criteria are: no occurrence of a periapical rarefaction in the furcation area; reduction or maintenance of an already present bone rarefaction in the furcation area of posterior teeth, maintaining the periradicular space, root resorption compatible with the eruptive phase and absence of pathological bone resorption. To evaluate the reduction of lesions or appearance of new lesions, we will compare the initial and final radiographs.
  Despite the anticipated time frame of 1 year, some participants were evaluated after this period due to the pandemic. The follow-up periods were until 24 months, and the final analysis were adjusted for this protocol deviation.

SECONDARY OUTCOMES:
Post-operative fistula | 7 days
  Report of fistula or presence of pus on the area of the endodontic treatment. This variable was recorded through a phone call to the children's guardians, who answered if they had noticed any purulent secretion in the area of the endodontically treated tooth (yes or no - dichotomous variable).
Post-operative pain | 7 days
  Report of post-operative pain until 7 days after the procedure. This outcome was collected through a phone call with the children's guardians, who asked if their child had reported any pain in the area of the procedure and if the participant had taken an analgesic (yes or no - dichotomous variable).
Post-operatve oedema | 7 days
  Report of post-operative oedema on the area of the endodontic treatment. This variable was recorded through a phone call to the children's guardians, who answered if they had noticed any oedema or swelling in the area of the endodontically treated tooth (yes or no - dichotomous variable).
Quality of root canal filling | Imediatelly after the treatment
  This variable was evaluated in the radiographs taken immediately after the endodontic treatment. An external observer, blinded to the allocated group, classified the quality of the root canal filling in adequate (filling to within 1 mm of the radiographic apex), before the apex (more than 1 mm of the radiographic apex) or with filling material overflow. This is a nominal qualitative variable (3 categories).

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No